CLINICAL TRIAL: NCT02373670
Title: Parent Mentors Using Positive Deviance in Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-470H
Record Dates: First submitted 2015-02-20; First posted 2015-02-27 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Obesity
Keywords: Positive deviance; Peer mentors
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parent Mentor (Experimental): Parent mentors using positive deviance findings to promote healthy behaviors
  Interventions: Behavioral: Promotion of positive deviance behaviors
- Education (Active Comparator): Community health workers providing health education to promote healthy behaviors
  Interventions: Behavioral: Promotion of healthy behaviors

INTERVENTIONS:
Behavioral: Promotion of positive deviance behaviors — Using locally derived positive deviance findings to inform a behavioral intervention
  Arms: Parent Mentor
Behavioral: Promotion of healthy behaviors — Using standardized healthy behavior education (EatPlayGrow curriculum from NHLBI)
  Arms: Education

SUMMARY:
A feasibility study randomizing participants (parents of children age 2-5 years old) to receive either education or a parent mentor with the aim of improving health behaviors and improving their body mass index z-score.

ELIGIBILITY:
Inclusion Criteria:

* BMI z-score >2

Exclusion Criteria:

* Medical conditions or receiving medications affecting weight

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Body mass index z-score | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Derived] Hollister EB, Foster BA, Dahdouli M, Ramirez J, Lai Z. Characterization of the Stool Microbiome in Hispanic Preschool Children by Weight Status and Time. Child Obes. 2018 Feb/Mar;14(2):122-130. doi: 10.1089/chi.2017.0122. Epub 2017 Oct 13. PMID 29028448
- [Derived] Foster BA, Aquino CA, Gil M, Gelfond JA, Hale DE. A Pilot Study of Parent Mentors for Early Childhood Obesity. J Obes. 2016;2016:2609504. doi: 10.1155/2016/2609504. Epub 2016 Jun 9. PMID 27379182